CLINICAL TRIAL: NCT03578588
Title: Single-dose Pharmacokinetic, Multiple-dose Tolerability and Pharmacokinetic Studies of Benapenem for Injection in Phase I Clinical Healthy Subjects
Brief Title: Benapenem PK Phase Ib Multiple-dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5081-CPK-1002
Record Dates: First submitted 2018-05-17; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-05

CONDITIONS: Health, Subjective
Keywords: single dose; multiple dose; Pharmacokinetic; Tolerability; Healthy Subject; Benapenem

STUDY DESIGN:
Intervention Model Description: A single-center, randomized, open-label, three-period and three-crossover trial design is adopted in the single-dose pharmacokinetic study; A single-center, randomized, open- label, and dose escalation trial design is used in the multiple-dose tolerability and pharmacokinetic studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Banapenem B1 group (Experimental): Dose in the 1st period 250mg; Dose in the 2nd period 500mg; Dose in the 3rd period 1000mg
  Interventions: Drug: Banapenem
- Banapenem B2group (Experimental): Dose in the 1st period 500mg; Dose in the 2nd period 1000mg; Dose in the 3rd period 250mg
  Interventions: Drug: Banapenem
- Banapenem B3group (Experimental): Dose in the 1st period 1000mg; Dose in the 2nd period 250mg; Dose in the 3rd period 500mg
  Interventions: Drug: Banapenem
- Banapenem C1group (Experimental): 250mg Once daily for 7 consecutive days
  Interventions: Drug: Banapenem
- Banapenem C2group (Experimental): 500mg Once daily for 7 consecutive days
  Interventions: Drug: Banapenem

INTERVENTIONS:
Drug: Banapenem — Twelve healthy adult volunteers, half male and female, are enrolled and randomly assigned to three groups, B1, B2, and B3. The subjects in three groups receive three doses, 250 mg, 500 mg and 1000 mg. Each group of subjects receive single-dose test drug at different dosages in each period. The subjects are divided into two groups, C1 and C2, 12 subjects in each group, half males and half females. 250 mg group is performed first. After completion of observation and confirming that the drug can be safely tolerated, study on 500 mg group is then performed
  Other Names: 5081

SUMMARY:
A single-center, randomized, open-label, three-period and three-crossover trial design is adopted in the single-dose pharmacokinetic study. 12adult volunteers, are assigned to 3 groups, B1（250mg), B2 (500mg), and B3 (1000mg). Each group of subjects receive single-dose test drug at different dosages in each period.

The tolerability and pharmacokinetic studies are performed simultaneously. Two doses, 250 mg and 500 mg, are proposed for multiple-dose tolerability and pharmacokinetic studies. The subjects are divided into two groups, C1 and C2, 12 subjects in each group, half males and half females. 250 mg group is performed first. Each subject receives only one dose, intravenous drip, once daily, for 7 consecutive days

DETAILED DESCRIPTION:
A single-center, randomized, open-label, three-period and three-crossover trial design is adopted in the single-dose pharmacokinetic study. Twelve healthy adult volunteers, half male and female, are enrolled and randomly assigned to three groups, B1, B2, and B3. The subjects in three groups receive three doses, 250 mg, 500 mg and 1000 mg. Each group of subjects receive single-dose test drug at different dosages in each period.

A single-center, randomized, open- label, and dose escalation trial design is used in the multiple-dose tolerability and pharmacokinetic studies. The tolerability and pharmacokinetic studies are performed simultaneously. Two doses, 250 mg and 500 mg, are proposed for multiple-dose tolerability and pharmacokinetic studies. The subjects are divided into two groups, C1 and C2, 12 subjects in each group, half males and half females. 250 mg group is performed first. After completion of observation and confirming that the drug can be safely tolerated, study on 500 mg group is then performed. Each subject receives only one dose, intravenous drip, once daily, for 7 consecutive days

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy subjects, aged 18 ~ 45;
* Body weight ≥ 50 kg and body mass index 19.0 ~ 24.0 kg/m2;
* Prior to the test, physical examination, blood routine, urine routine, liver and kidney functions, and related examinations normal, or mild abnormalities in indicators while without clinical significance as indicated by the investigator
* Normal or mild abnormalities without clinical significance in the standard 12-lead ECG;
* Signing informed consent form

Exclusion Criteria:

* Regular smoking, alcohol abuse, and drug abuse;
* Use of drugs with known damage to an organ within three months;
* History of specific allergies, or history of drug allergy, especially those allergic to lactams and excipients of test drug;
* Febrile illnesses within three days before the screening;
* Patients with mental illness or psychotic disorder in the past;
* Past mental and nervous system diseases (epilepsy, stroke, cerebrovascular disorder, etc.), gastrointestinal disorder (such as stomach ulcers, gastritis, etc.) or disorder of other systems (such as cardiovascular, respiratory, hematological, or endocrine system, etc.) diseases or medical history.
* Taking any medication, including traditional Chinese medicine;
* Having taken any medication that may affect test results within two weeks before the screening, such as antibiotics, NSAIDs, aluminum- or magnesium-containing antacids, diuretics, anticoagulants, central nervous system depressants, and any drug that may affect the drug absorption;
* Having participated in other investigational drug trial in the preceding three months;
* Blood donation for 360 ml or more within three months before the screening;
* Heart rate<50 bpm or >100 bpm;
* Systolic blood pressure < 90 mmHg or ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg or < 60 mmHg;
* Women who are pregnant or breastfeeding, or who may be pregnant without adopting acceptable contraception, or who have a positive result in serum pregnancy test;
* Women who are planning to become pregnant within 6 months, or male subjects who are planning to make his spouse pregnant within 6 months;
* HBsAg, HCV antibody, HIV antibody, and Treponema Pallidum antibody positive;
* Urine drug-of-abuse testing positive;
* Any other factor that makes the subject not suitable for the trial as indicated by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2016-01-13 (Actual); Study Completion 2016-01-13 (Actual)

PRIMARY OUTCOMES:
AUC(0-24) of Benapenem | Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24,36,48 hours after Dosing
  AUC(0-24) is the area under the curve from time 0 to 24 hours
Maximum observed plasma concentration (Cmax) of Benapenem | Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24,36,48 hours after Dosing
  Maximum observed plasma concentration (Cmax) of following in healthy subjects
Time to maximum observed plasma concentration (tmax) of Benapenem | Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24,36,48 hours after Dosing
  Time to maximum observed plasma concentration (tmax)
Time to elimination half-life (t1/2) of Benapenem | Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 3, 4, 6,8,12, 24,36,48 hours after Dosing
  Time to elimination half-life (t1/2)

SECONDARY OUTCOMES:
Number of subjects with clinically significant findings in vital signs | Screening and Day1, Day 2, Day4 after dosing
  Vitals signs such as systolic and diastolic blood pressure, heart rate, and pulse rate will be measured in a semi-supine position after 5 minutes of rest
Number of subjects with clinically significant findings in laboratory parameters | Screening and Day1, Day 2, Day4 after dosing
  Hematology and Clinical Chemistry and Urine routine abnormalities will be monitored
Number of subjects with adverse events and serious adverse events | Screening and Day1, Day 2, Day4 after dosing
Number of subjects with clinically significant 12-lead ECGs | Screening and Day1, Day 2, Day4 after dosing
  Single 12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, and QT intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Lv, PhD, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data to other researchers.

REFERENCES:
- [Derived] Zhao CY, Lv Y, Zhu Y, Wei MJ, Liu MY, Ji XW, Kang ZS, Xia YH, Tian JH, Ma Y, Liu Y. A First-in-Human Safety, Tolerability, and Pharmacokinetics Study of Benapenem in Healthy Chinese Volunteers. Antimicrob Agents Chemother. 2019 Feb 26;63(3):e02188-18. doi: 10.1128/AAC.02188-18. Print 2019 Mar. PMID 30617093